CLINICAL TRIAL: NCT07407348
Title: Bioequivalence of Two Survodutide (BI 456906) Formulations Via Subcutaneous Administration After Multiple Doses (an Open-label, Randomised, Multiple-dose, Crossover Trial)
Brief Title: A Study in People With Overweight or Obesity to Compare How 2 Different Formulations of Survodutide Are Taken up by the Body
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1404-0066; U1111-1323-8960 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formulation A, then Formulation B6 (Experimental)
  Interventions: Combination Product: Formulation A; Combination Product: Formulation B6
- Formulation B6, then Formulation A (Experimental)
  Interventions: Combination Product: Formulation A; Combination Product: Formulation B6

INTERVENTIONS:
Combination Product: Formulation A — Formulation A of survodutide
Combination Product: Formulation B6 — Formulation B6 of survodutide

SUMMARY:
The primary objective of this trial is to assess bioequivalence of two formulations of survodutide (formulation A and formulation B6) after multiple-dose treatment in male and female trial participants living with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female trial participant according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 65 years (inclusive)
3. Body Mass Index (BMI) of 27.0 to 39.9 Kg/ m^2 (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
5. For women of child-bearing potential (WOCBP) trial participants: Woman of childbearing potential (WOCBP) trial participants who meet any of the following criteria for a highly effective contraception from at least 28 days before the first administration of trial medication until 28 days after trial completion:

   * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal). In case of oral contraception, a barrier method should be used in addition or advised to change to non-oral contraceptives at least 7 days prior to first dose of investigational medicine product (IMP)
   * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants). In case of oral contraception, a barrier method should be used in addition or advised to change to non-oral contraceptives at least 7 days prior to first dose of IMP
   * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
   * Complete abstinence (refraining from heterosexual intercourse during the entire period of risk associated with the study treatment) is considered a highly effective method of contraception only if it is in line with the preferred and usual lifestyle of the trial participant. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to trial IMP, spermicides only, lactational amenorrhoea method (LAM) and withdrawal are not acceptable methods of contraception
   * Bilateral tubal ligation/occlusion is considered a highly effective method of contraception, provided that the procedure has not been reversed or failed.
   * Surgically sterilised (including hysterectomy, bilateral salpingectomy and bilateral oophorectomy)
   * Postmenopausal, defined as no menses for 1 year without an alternative medical cause

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR) or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic Blood pressure (BP) outside the range of 90 to 150 mmHg, diastolic BP outside the range of 50 to 100 mmHg, or PR outside the range of 50 to 100 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
6. Diseases of the Central nervous system (CNS) (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
7. History of relevant orthostatic hypotension, fainting spells, or blackouts
8. Relevant chronic or acute infections within the 4 weeks prior to screening Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-01-26 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve of survodutide in plasma at steady state over a uniform dosing interval tau (AUC tau,ss) | Up to 239 days.
Maximum measured concentration of survodutide in plasma at steady state over a uniform dosing interval tau (Cmax,ss) | Up to 239 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency